CLINICAL TRIAL: NCT01582711
Title: TBTC Study 33. An Evaluation of Adherence to Latent Tuberculosis Infection (LTBI) Treatment With 12 Doses of Once Weekly Rifapentine (RPT) and Isoniazid (INH) Given as Self-administered (SAT) Versus Directly-observed Therapy (DOT): iAdhere.
Brief Title: Study 33: Adherence to Latent Tuberculosis Infection Treatment 3HP SAT Versus 3HP DOT
Acronym: iAdhere
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP 6222; TBTC Study 33 (Other: CDC)
Record Dates: First submitted 2012-02-10; First posted 2012-04-23 (Estimated); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Latent Tuberculosis Infection
Keywords: LTBI; LTB; Latent TB; TB infection
MeSH Terms: conditions — Latent Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3HP Directly Observed Therapy (DOT) (Active Comparator): 900mg of isoniazid plus 900mg of rifapentine given weekly for 3 months (12 weeks, 12 doses) under Directly Observed Therapy (DOT)
  Interventions: Drug: isoniazid and rifapentine
- 3HP Self Administered Therapy (SAT) (Experimental): 900mg of isoniazid plus 900mg of rifapentine given weekly for 3 months (12 weeks, 12 doses) as patient Self Administered Therapy (SAT)
  Interventions: Behavioral: Self Administered Therapy (SAT); Drug: isoniazid and rifapentine
- 3HP SAT with SMS Reminders (Experimental): 900mg of isoniazid plus 900mg of rifapentine given weekly for 3 months (12 weeks, 12 doses) as patient Self Administered Therapy (SAT). In addition, patient receives phone Short Message Service (SMS) reminders weekly.
  Interventions: Behavioral: Self Administered Therapy (SAT); Behavioral: SMS reminders; Drug: isoniazid and rifapentine

INTERVENTIONS:
Behavioral: Self Administered Therapy (SAT) — Self Administered Therapy (SAT)
  Other Names: SAT
  Arms: 3HP SAT with SMS Reminders; 3HP Self Administered Therapy (SAT)
Behavioral: SMS reminders — Short Message Service (SMS) text reminders
  Other Names: SMS; phone text reminder
  Arms: 3HP SAT with SMS Reminders
Drug: isoniazid and rifapentine — rifapentine (PRIFTIN, RPT) 900 mg and isoniazid (INH) 900mg, once-weekly, for 12 weeks (12 doses)
  Other Names: PRIFTIN; RPT; P; INH; I

SUMMARY:
The study is an open label, multicenter, randomized (three arms: DOT (standard control), SAT, SAT with SMS reminders) controlled clinical trial. The trial is conducted in patients diagnosed with latent tuberculosis infection (LTBI) who are recommended for treatment. The primary objective is to evaluate adherence to a three-month (12-dose) regimen of weekly rifapentine and isoniazid (3RPT/INH) given by directly observed therapy (DOT) compared to self-administered therapy (SAT). The secondary objectives:

* To compare the treatment completion rates between participants randomized to SAT without reminders versus SAT with weekly SMS reminders
* To evaluate the timing of doses and patterns of adherence to once weekly RPT/INH among participants who complete treatment and those who discontinue therapy prior to completion.
* To determine the availability and acceptability of using SMS reminders among all patients consenting to participate in the study.
* To determine the toxicity and tolerability by comparing the rates of any drug-related grade 3 or 4 adverse events or death between the DOT arm and the SAT arms (both combined and individually)
* To compare the frequency, timing, and causes for failure to complete treatment between the DOT arm and the SAT arms
* To collect patient-specific cost data related to the 3 treatment arms
* To describe the pattern of antituberculosis drug resistance among Mycobacterium tuberculosis strains cultured from participants who develop active TB.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that approximately 2.3 billion people are infected with Mycobacterium tuberculosis. Approximately 1.7 million people die of TB each year, the second most common infectious cause of death in the world. In order to improve TB control worldwide, an affordable, effective, short course treatment for latent TB infection (LTBI) is a global priority.

Candidates for LTBI treatment are those persons with a positive TST or IGRA, particularly if they also have risk factors for progressing to active TB, including individuals likely to be recently infected. The Prevent TB Study (TBTC Study 26) was an open-label, randomized, phase III controlled clinical trial with over 8,000 high risk TST reactors enrolled. The study compared rifapentine and INH (3RPT/INH) given once-weekly by directly observed treatment (DOT) for 3 months (12 doses) compared with 9 months of daily, self-administered INH. The results demonstrated the safety and efficacy of the shorter regimen. Moreover, the once weekly therapy had significantly higher treatment completion rates than the standard 9 INH regimen.

One of the most effective strategies for assuring adherence with therapy is to have each dose of medication directly administered by a health care worker who observes and records the ingestion of the drugs. DOT for active TB has been successfully used in many settings to improve treatment completion, however cost and logistical constraints of DOT remain. The estimated cost of giving 12 weekly DOT doses to all LTBI patients is likely prohibitive for TB control programs worldwide. This may lead to a decreased uptake of the new regimen or implementation using SAT where adherence has not been studied. Therefore, to apply the Prevent TB study results more broadly, a new study evaluating treatment completion of 3 RPT/INH given as SAT is conducted.

Medication adherence is defined by whether patients take a treatment as prescribed. The effectiveness of any treatment is determined largely by adherence. In clinical practice and research, indirect measures of adherence are commonly used. Indirect measures of adherence include patient self-report, evaluation of pharmacy dispensation records, pill counts, and the use of electronic prescription bottle monitors. Patient self-reported adherence is accurate when non-adherence is reported but tends to overestimate true adherence. Self-report is not discerning enough to be utilized as a sole measure of adherence in research settings where adherence is the primary outcome. Pill counts have been utilized successfully in research and clinical settings for real-time assessment but also tend to overestimate adherence. Electronic drug monitors such as the Medication Event Monitoring System (MEMS) are the best available tools to assess the timing and patterns of adherence. This study uses a combination of indirect measures including MEMS, pill counts, and self-report to provide the most accurate assessment of adherence to once weekly, self-administered RPT/INH.

The number of cellular phone users globally has increased dramatically in the last decade. Cell phones and SMS reminders have been used successfully in randomized controlled clinical trials to improve adherence to vaccines, HIV medications, and asthma treatment. SMS appear to be cost-effective ways to reach patients in remote locations. This study examines effect of SMS on medication adherence.

The goal of this open label clinical trial is to compare the adherence to 3RPT/INH given by DOT versus SAT or SAT with a weekly SMS reminder. The primary assessment of adherence will be treatment completion which is defined as taking at least 90% of the doses (11/12 doses of each drug) within 16 weeks of initiation. Secondary objectives include evaluating the patterns of adherence in participants who fail to complete, determining the feasibility and impact of using SMS reminders on treatment completion with SAT, evaluating the tolerability and any adverse events associated with each treatment arm, monitoring for the development of active TB, determining the drug susceptibility for participants who develop active TB, and measuring important patient-related expenditures associated with each study arm. The trial will be conducted in patients diagnosed with LTBI and recommended for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-nursing females
* Age > 18 years
* Weight > 45kg and considered appropriate to receive RPT 900mg and INH 900mg once weekly by the local site investigator
* Willingness to provide signed informed consent.
* Clinical indication for LTBI treatment such as: 1) persons with a positive tuberculin skin test (TST) as defined by CDC criteria or a positive interferon-gamma release assay (IGRA) defined per the manufacturers' guidelines AND one of the following: close contact to someone with culture confirmed TB, HIV infection, or > 2 cm2 of pulmonary parenchymal fibrosis on chest X-ray and no prior history of TB treatment; 2) TST or IGRA converters defined as a documented change from negative to positive within a two-year period; 3) Persons with any other clinical indication for LTBI treatment as locally defined including persons with a negative TST and/or IGRA (e.g. HIV-infected close contacts to an active pulmonary TB cases)

Exclusion Criteria:

* Confirmed or suspected active TB
* Contacts to a source case with known resistance to isoniazid or rifampin
* Persons with a history (by written documentation or self-report) of ever receiving > 1 week of treatment for active or latent TB, regardless of whether the course was completed, because adherence may be different in people who previously took TB treatment
* Persons who are not considered candidates for SAT by the local investigator
* History of sensitivity or intolerance to isoniazid or rifamycins
* Serum alanine aminotransferase (ALT, SGPT) > 5x upper limit of normal among persons in whom an ALT is determined
* Persons with HIV-infection who 1) have a CD4 < 350 or 2) are currently receiving or planning to receive antiretroviral therapy in the first 120 days after study initiation (e.g., HIV-1 protease inhibitors, nucleoside or non-nucleoside reverse transcriptase inhibitors, CCR5 inhibitors or integrase inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey S Borisov, MD, MPH, Study Director — U.S. Centers for Disease Control and Prevention (CDC), Atlanta, USA.; Robert Belknap, MD, Study Chair — Division of Infectious Diseases, University of Colorado, Denver, USA.; Robert Belknap, MD, Principal Investigator — Division of Infectious Diseases, University of Colorado, Denver, USA.
Locations (12):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Denver Public Health Department, Denver, Colorado
  - Washington DC Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - Columbia University College of Physicians and Surgeons and New York City Department of Health, New York, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center and Nashville Metro Public Health Department, Nashville, Tennessee
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - South Texas - Department of State Health Services, San Antonio, Texas
- TB and Chest service of Hong Kong, Hong Kong, China
- Wits Health Consortium, Soweto, South Africa
- Agencia de Salut Publica - Barcelona, Spain and UNTHSC, Barcelona, Spain

REFERENCES:
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Centers for Disease Control and Prevention (CDC). Recommendations for use of an isoniazid-rifapentine regimen with direct observation to treat latent Mycobacterium tuberculosis infection. MMWR Morb Mortal Wkly Rep. 2011 Dec 9;60(48):1650-3. PMID 22157884
- [Background] Shepardson D, Marks SM, Chesson H, Kerrigan A, Holland DP, Scott N, Tian X, Borisov AS, Shang N, Heilig CM, Sterling TR, Villarino ME, Mac Kenzie WR. Cost-effectiveness of a 12-dose regimen for treating latent tuberculous infection in the United States. Int J Tuberc Lung Dis. 2013 Dec;17(12):1531-7. doi: 10.5588/ijtld.13.0423. PMID 24200264
- [Background] Sterling TR, Moro RN, Borisov AS, Phillips E, Shepherd G, Adkinson NF, Weis S, Ho C, Villarino ME; Tuberculosis Trials Consortium. Flu-like and Other Systemic Drug Reactions Among Persons Receiving Weekly Rifapentine Plus Isoniazid or Daily Isoniazid for Treatment of Latent Tuberculosis Infection in the PREVENT Tuberculosis Study. Clin Infect Dis. 2015 Aug 15;61(4):527-35. doi: 10.1093/cid/civ323. Epub 2015 Apr 22. PMID 25904367
- [Derived] Sadowski C, Belknap R, Holland DP, Moro RN, Chen MP, Wright A, Millet JP, Cayla JA, Scott NA, Borisov A, Gandhi NR. Symptoms and Systemic Drug Reactions in Persons Receiving Weekly Rifapentine Plus Isoniazid (3HP) Treatment for Latent Tuberculosis Infection. Clin Infect Dis. 2023 Jun 16;76(12):2090-2097. doi: 10.1093/cid/ciad083. PMID 36815322
- [Derived] Moro RN, Scott NA, Vernon A, Tepper NK, Goldberg SV, Schwartzman K, Leung CC, Schluger NW, Belknap RW, Chaisson RE, Narita M, Machado ES, Lopez M, Sanchez J, Villarino ME, Sterling TR. Exposure to Latent Tuberculosis Treatment during Pregnancy. The PREVENT TB and the iAdhere Trials. Ann Am Thorac Soc. 2018 May;15(5):570-580. doi: 10.1513/AnnalsATS.201704-326OC. PMID 29393655
- [Derived] Belknap R, Holland D, Feng PJ, Millet JP, Cayla JA, Martinson NA, Wright A, Chen MP, Moro RN, Scott NA, Arevalo B, Miro JM, Villarino ME, Weiner M, Borisov AS; TB Trials Consortium iAdhere Study Team. Self-administered Versus Directly Observed Once-Weekly Isoniazid and Rifapentine Treatment of Latent Tuberculosis Infection: A Randomized Trial. Ann Intern Med. 2017 Nov 21;167(10):689-697. doi: 10.7326/M17-1150. Epub 2017 Nov 7. PMID 29114781
- See also: Home page of the Tuberculosis Trials Consortium (TBTC) funded by the U.S. Centers for Disease Control and Prevention (CDC) — https://www.cdc.gov/tb/research/tbtc.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Started | 337 | 337 | 328
Completed | 337 | 337 | 328
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders | Total
Number analyzed (Participants) | 337 | 337 | 328 | 1002
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [27 to 48] | 36 [27 to 48] | 38 [27 to 49] | 36 [27 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 161 | 168 | 482
  Male | 184 | 176 | 160 | 520
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 68 | 62 | 70 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 84 | 91 | 75 | 250
  White | 171 | 175 | 172 | 518
  More than one race | 14 | 9 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 261 | 262 | 251 | 774
  China | 15 | 14 | 16 | 45
  South Africa | 26 | 29 | 28 | 83
  Spain | 35 | 32 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion Rate.
Description: To compare the treatment completion rates between participants randomized to DOT vs SAT without reminders and DOT versus SAT with weekly SMS reminders. Treatment completion is defined as taking at least 90% of the doses (11/12 doses of each drug) within 16 weeks of treatment initiation.
Time Frame: Up to 16 weeks from start of treatment.
Population: Participants analyzed excludes 4 participants (2 in each SAT groups) who were enrolled as contacts of a person with active TB before susceptibility results had returned showing resistance to isoniazid or rifampin in source patient. These participants were excluded from treatment completion analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 337 | 335 | 326
Participants | 294 | 248 | 250

2. Secondary Outcome: Treatment Completion Rates Between Participants Randomized to SAT Without Reminders Versus SAT With Weekly SMS Reminders
Description: To compare the treatment completion rates between participants randomized to SAT without reminders versus SAT with weekly SMS reminders
Time Frame: Up to 16 weeks from start of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 335 | 326
Participants | 248 | 250

3. Secondary Outcome: The Percentage of Participants Who Completed Treatment Based on SOC vs SOC Plus MEMS
Description: The number and proportion of participants who adhered (completed treatment) based on pill count and self-report, considered to be standard of care (SOC) vs. the number of participants who completed treatment based on SOC plus MEMS cap.
Time Frame: Up to 16 weeks from start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 337 | 337 | 328
Participants
  Treatment completion proportion based on pill count/self-report | 294 | 271 | 266
  Treatment completion proportion based on pill count/self-report and MEMS cap | 294 | 248 | 249

4. Secondary Outcome: Availability and Acceptability
Description: To determine the availability and acceptability of using SMS reminders among all patients consenting to participate in the study.
Time Frame: Up to 16 weeks from start of treatment.
Population: 'Proportion of Participants willing to use SMS (Acceptability) (eSAT arm ONLY)' analysis was only done in '3HP SAT with SMS Reminders'.
Measure: Count of Participants; unit: Participants
Groups:
- 3HP Directly Observed Therapy (DOT): 900mg of isoniazid plus 900mg of rifapentine given weekly for 3 months (12 weeks, 12 doses) under Directly Observed Therapy (DOT) isoniazid and rifapentine: rifapentine (PRIFTIN, RPT) 900 mg and isoniazid (INH) 900mg, once-weekly, for 12 weeks (12 doses)
Arm/Group | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders | 3HP Directly Observed Therapy (DOT)
Number analyzed (Participants) | 337 | 328 | 337
Participants
  Proportion of Participants have cell SMS phone (Availability) | 34 | 29 | 28
  Proportion of Participants willing to use SMS (Acceptability) (eSAT arm ONLY): number analyzed (Participants) | 0 | 328 | 0
  Proportion of Participants willing to use SMS (Acceptability) (eSAT arm ONLY) | 0 | 229 | 0

5. Secondary Outcome: Number and Percentage of Participants With Drug-related Grade 3 or 4 Adverse Events or Death
Description: To determine the toxicity and tolerability by comparing the rates of any drug-related grade 3 or 4 adverse events or death between the DOT arm and the SAT arms (both combined and individually)
Time Frame: Up to 16 weeks from start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 337 | 337 | 328
Participants | 23 | 23 | 29

6. Secondary Outcome: Number and Percentage of Participants Reason for Failure to Complete Treatment
Description: To compare the frequency, timing, and causes for failure to complete treatment between the DOT arm and the SAT arms (both combined and individually) including discontinuation due to:
  * non-adherence
  * any adverse event (AE)
  * a diagnosis of active TB
  * other reasons
Time Frame: Up to 16 weeks from start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 337 | 337 | 328
Participants
  Study therapy not started | 3 | 7 | 4
  Drug toxicities causing permanent discontinuation | 12 | 18 | 14
  Failure to complete minimum number of PP doses | 4 | 7 | 9
  Not advisable to continue study drugs | 2 | 5 | 2
  Refused further study therapy | 6 | 7 | 11
  Patient became pregnant | 2 | 1 | 2
  Other | 9 | 12 | 11
  Unknown/Missing | 2 | 6 | 6

7. Secondary Outcome: Patient-specific Cost
Description: To collect patient-specific cost data related to the DOT and SAT arms
Time Frame: Up to 20 weeks from start of treatment.
Population: This analysis was conducted in 81 (DOT-40, SAT-41) participants from 7 study sites. As pre-specified in the protocol, DOT cost maybe prohibitive to TB programs, and SAT cost may provide a cost-effective alternative. Data was collected and analyzed to assess DOT costs vs SAT costs, such that the distinction between SAT and eSAT arms were not appropriate. As a result, participants in the SAT arms were combined to find total cost.
Measure: Median (Inter-Quartile Range); unit: U.S. Dollar
Groups:
- 3HP Self Administered Therapy (Combined SAT and SAT With Reminders): 900mg of isoniazid plus 900mg of rifapentine given weekly for 3 months (12 weeks, 12 doses) as patient Self Administered Therapy (SAT)
  Self Administered Therapy (SAT): Self Administered Therapy (SAT)
  isoniazid and rifapentine: rifapentine (PRIFTIN, RPT) 900 mg and isoniazid (INH) 900mg, once-weekly, for 12 weeks (12 doses)
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (Combined SAT and SAT With Reminders)
Number analyzed (Participants) | 40 | 41
U.S. Dollar | 361.50 [125 to 425] | 257.82 [90 to 340]

8. Secondary Outcome: Antituberculosis Drug Resistance
Description: To describe the pattern of antituberculosis drug resistance among Mycobacterium tuberculosis strains cultured from participants who develop active TB.
Time Frame: Up to 16 weeks from start of treatment.
Population: Participants analyzed excludes 4 participants (2 in each SAT groups) who were enrolled as contacts of a person with active TB before susceptibility results had returned showing resistance to isoniazid or rifampin in source patient. These participants were excluded from drug resistance analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
Number analyzed (Participants) | 337 | 335 | 326
Participants
  Developed TB but not drug resistant | 0 | 0 | 1
  Antituberculosis Drug Resistant | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of study treatment (up to 16 weeks) + 14 days (for late toxicity)
Arm/Group | 3HP Directly Observed Therapy (DOT) | 3HP Self Administered Therapy (SAT) | 3HP SAT With SMS Reminders
All-Cause Mortality (participants affected / at risk) | 0/337 | 0/337 | 1/328
Serious Adverse Events (participants affected / at risk) | 11/337 | 5/337 | 6/328
Other Adverse Events (participants affected / at risk) | 42/337 | 54/337 | 56/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3HP Directly Observed Therapy (DOT) (N=337) | 3HP Self Administered Therapy (SAT) (N=337) | 3HP SAT With SMS Reminders (N=328)
Acute gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Systemic Drug Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
rheumatoid arthritis flare (General disorders) | 1 (1) | 0 (0) | 0 (0) — related to reduced efficacy of prednisone due to rifapentine
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
unrelated to study drug (General disorders) | 8 (8) | 5 (5) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3HP Directly Observed Therapy (DOT) (N=337) | 3HP Self Administered Therapy (SAT) (N=337) | 3HP SAT With SMS Reminders (N=328)
Systemic Drug Reaction (General disorders) | 13 (13) | 15 (15) | 14 (14)
Hepatitis (General disorders) | 1 (1) | 3 (3) | 5 (5)
Thrombocytopenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Other (General disorders) | 27 (27) | 36 (36) | 50 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No